CLINICAL TRIAL: NCT03962894
Title: Early Administration of Steroids in the Ambulance Setting: An Observational Design Trial
Brief Title: Early Administration of Steroids in the Ambulance Setting
Acronym: EASI-AS-ODT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201901351 -N-A; 1K23HL149991-01 (NIH)
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Prehospital Systemic Corticosteroids (Experimental): Children with asthma attacks who receive systemic corticosteroids in the prehospital environment by emergency medical services
  Interventions: Drug: Prednisolone
- Usual Care (No Intervention): Children with asthma attacks treated by emergency medical services who receive usual care en route to emergency departments, where in the ED they then receive systemic corticosteroids

INTERVENTIONS:
Drug: Prednisolone — During a sequenced rollout protocol change for several EMS agencies, those agencies will adopt protocol change to administer prednisolone to children with asthma attacks in the prehospital environment prior to ED arrival.
  Arms: Early Prehospital Systemic Corticosteroids

SUMMARY:
Asthma is the most common chronic disease of childhood and is a leading cause of emergency medical treatment. For children experiencing an asthma exacerbation, emergency department (ED) guidelines recommend early systemic corticosteroid (CS) administration, since studies have shown associated, time-sensitive, decreases in hospital admissions and ED length-of-stay (LOS). For patients who are treated by 911 emergency medical services (EMS) first, there exists an opportunity for even earlier administration of CS, prior to ED arrival. Yet, preliminary data demonstrate that currently less than 10% of EMS pediatric asthma patients receive CS prior to ED arrival.

Given the known time-sensitivity of CS' effects on patient outcomes, the investigators hypothesize that even earlier EMS administration of CS will decrease hospital admissions, ED LOS, and intensive care unit admissions for pediatric patients with an acute asthma exacerbation. Using a pragmatic observation design in multiple EMS agencies, we will enroll patients to analyze clinical outcomes and comparative costs of EMS CS administration, and how both are influenced by EMS transport time. That novel combination of analyses will help build evidence-based guidelines adaptable for diverse EMS agencies nationwide.

ELIGIBILITY:
Inclusion Criteria:

* primary problem: Asthma exacerbation
* stable to take an oral medication
* transported by EMS to an ED

Exclusion Criteria:

* unconscious, hemodynamically unstable, or critically ill -> EMS will proceed with usual critical care (includes IV methylprednisolone as per protocol)
* daily or every other day corticosteroid therapy
* allergy to prednisolone or another corticosteroid
* chronic lung disease besides asthma, airway anatomic abnormalities, tracheostomy, immunocompromised, traumatic injury, pregnancy, law enforcement custody, non-English speaking

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 834 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fishe, MD, Principal Investigator — University of Florida
Locations (7):
- United States (7):
  - Walton County EMS, DeFuniak Springs, Florida
  - Lee County Public Safety & Emergency Services, Fort Myers, Florida
  - Sarasota County EMS, Sarasota, Florida
  - Leon County EMS, Tallahassee, Florida
  - Nassau County Fire Rescue Department, Yulee, Florida
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Texas Children's Hospital / UT Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was no recruitment, as this was an observational study of patients who were receiving EMS treatment regardless of the study.
Pre-assignment Details: EMS agencies who decided to incorporate oral systemic corticosteroids as part of clinical care were for this study. The study assigned the start date for EMS agencies to include oral systemic corticosteroids. For the purpose of analysis, we treated that as a stepped wedge protocol design. All agencies contributed one year of data for early prehospital systemic corticosteroids, and one year of data for no prehospital systemic corticosteroids.
Units Other Than Participants: EMS agencies
Groups:
- Houston EMS Pre and Post-Protocol Change: Children with asthma attacks treated by Houston EMS. Data abstracted 12 months before and 12 months after protocol change adding oral systemic corticosteroids that occurred on 10/1/2014.
- Cincinnati EMS Pre- and Post-Protocol Change: Children with asthma attacks treated by Cincinnati EMS. Data abstracted 12 months before and 12 months after protocol change adding oral systemic corticosteroids that occurred on 1/1/2016.
- Nassau County FL EMS Pre- and Post- Protocol Change: Children with asthma attacks treated by Nassau County FL EMS. Data abstracted 12 months before and 12 months after protocol change adding oral systemic corticosteroids that occurred on 6/1/2019.
- Lee County FL EMS Pre- and Post- Protocol Change: Children with asthma attacks treated by Lee County FL EMS. Data abstracted 12 months before and 12 months after protocol change adding oral systemic corticosteroids that occurred on 11/1/2019.
- Walton County FL EMS Pre- and Post-Protocol Change: Children with asthma attacks treated by Walton County FL EMS. Data abstracted 12 months before and 12 months after protocol change adding oral systemic corticosteroids that occurred on 11/1/2020.
- Leon County FL EMS Pre- and Post-Protocol Change: Children with asthma attacks treated by Leon County FL EMS. Data abstracted 12 months before and 12 months after protocol change adding oral systemic corticosteroids that occurred on 2/1/2021.
- Sarasota County FL EMS Pre- and Post-Protocol Change: Children with asthma attacks treated by Sarasota County FL EMS. Data abstracted 12 months before and 12 months after protocol change adding oral systemic corticosteroids that occurred on 6/1/2021/
Period: Overall Study
Arm/Group | Houston EMS Pre and Post-Protocol Change | Cincinnati EMS Pre- and Post-Protocol Change | Nassau County FL EMS Pre- and Post- Protocol Change | Lee County FL EMS Pre- and Post- Protocol Change | Walton County FL EMS Pre- and Post-Protocol Change | Leon County FL EMS Pre- and Post-Protocol Change | Sarasota County FL EMS Pre- and Post-Protocol Change
Started | 265; 1 EMS agencies (Data was abstracted for 12 months after each EMS agency adopted a protocol incorporating oral systemic corticosteroids in addition to IV systemic corticosteroids.) | 271; 1 EMS agencies | 6; 1 EMS agencies | 133; 1 EMS agencies | 14; 1 EMS agencies | 99; 1 EMS agencies | 46; 1 EMS agencies
Completed | 265; 1 EMS agencies (Data was abstracted for 12 months after each EMS agency adopted a protocol incorporating oral systemic corticosteroids in addition to IV systemic corticosteroids.) | 271; 1 EMS agencies | 6; 1 EMS agencies | 133; 1 EMS agencies | 14; 1 EMS agencies | 99; 1 EMS agencies | 46; 1 EMS agencies
Not Completed | 0; 0 EMS agencies | 0; 0 EMS agencies | 0; 0 EMS agencies | 0; 0 EMS agencies | 0; 0 EMS agencies | 0; 0 EMS agencies | 0; 0 EMS agencies

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Prehospital Systemic Corticosteroids | Usual Care | Total
Number analyzed (Participants) | 175 | 659 | 834
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8 [5 to 13] | 8 [5 to 12] | 8 [5 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 381 | 448
  Male | 108 | 278 | 386
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 107 | 417 | 524
  White | 37 | 146 | 183
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 92 | 121
Bronchodilator Administered [Count of Participants; unit: Participants] — Bronchodilators included albuterol and xopenex, administered either via inhaler or nebulizer
  Participants | 159 | 529 | 688

OUTCOME MEASURES:

1. Primary Outcome: Hospital Admission
Description: Number of admissions to an inpatient unit (general or ICU) for an asthma exacerbation
Time Frame: Day 1 (ED stay)
Measure: Count of Participants; unit: Participants
Groups:
- Early Prehospital Systemic Corticosteroids: Children with asthma attacks who receive systemic corticosteroids and bronchodilators in the prehospital environment by emergency medical services
- No Early Prehospital Systemic Corticosteroids: Children with asthma attacks treated by emergency medical services who receive bronchodilators en route to emergency departments, where in the ED they then receive systemic corticosteroids
Arm/Group | Early Prehospital Systemic Corticosteroids | No Early Prehospital Systemic Corticosteroids
Number analyzed (Participants) | 175 | 659
Participants | 57 | 208

2. Secondary Outcome: Emergency Department Length-of-stay
Description: Length of time in emergency department for patients from arrival to disposition (i.e., length of time for discharge, admission, or transfer to another hospital)
Time Frame: Day 1 (from EMS arrival to ED disposition)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Early Prehospital Systemic Corticosteroids | No Early Prehospital Systemic Corticosteroids
Number analyzed (Participants) | 175 | 659
minutes | 168 [127 to 256] | 159 [108 to 228]

ADVERSE EVENTS:
Time Frame: 2 years
Description: There were no serious AEs, no mortality, and no other non serious AEs observed in the study.
Arm/Group | Early Prehospital Systemic Corticosteroids | No Early Prehospital Systemic Corticosteroids
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/659
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/659
Other Adverse Events (participants affected / at risk) | 0/175 | 0/659

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT03962894/Prot_SAP_000.pdf